CLINICAL TRIAL: NCT05168995
Title: Effects of Beclometasone Dipropionate/Formoterol Fumarate Fixed Combination Administered With the NEXT(Haler) in a Real-world Study on the Probability of Improving the Asthma Control Status After 6 Months of Treatment. The NEWTON Study
Brief Title: Effects of Beclometasone Dipropionate/Formoterol Fumarate Via NEXT(Haler) in a Real-world Study on Asthma Control
Acronym: NEWTON
Status: Completed | Type: Observational
Sponsor: Chiesi Italia (Industry)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Other Study IDs: CHIT-2101
Record Dates: First submitted 2021-12-10; First posted 2021-12-23 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Asthma
Keywords: Control; PROs
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthmatic patients in treatment with BDP/FF NEXThaler® 100/6 micrograms: Not adequately controlled asthmatic patients in treatment with Beclometasone dipropionate (BDP)/formoterol fumarate (FF) 100/6 micrograms per actuation inhalation powder via NEXThaler®
  Interventions: Drug: BDP/FF NEXThaler® 100/6 micrograms

INTERVENTIONS:
Drug: BDP/FF NEXThaler® 100/6 micrograms — BDP/FF NEXThaler® 100/6 maintenance treatment: one or two inhalations twice daily (one inhalation in the morning and one inhalation in the evening).
  BDP/FF NEXThaler® 100/6 maintenance and reliever treatment (MART)

SUMMARY:
The goal of asthma management is to achieve and maintain optimal asthma control. The NEWTON study assesses the evolution over time of patient reported outcomes (PROs) in asthmatic patients, not adequately controlled with ongoing treatments and initiating therapy with extrafine beclometasone dipropionate/formoterol fumarate (BDP/FF) via NEXThaler.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years;
2. Patients enrolled on the same day as the first prescription with BDP/FF NEXThaler® 100/6 micrograms, or having ongoing treatment with BDP/FF NEXThaler® 100/6 micrograms started within the previous 14 days (maximum), as per local standard clinical practice.
3. Not adequately controlled asthmatic patients (according to clinician's judgement) when BDP/FF NEXThaler® 100/6 micrograms was prescribed;
4. Patients not treated with extrafine formulations during the 6 months before starting the treatment with BDP/FF NEXThaler®;
5. Written informed consent to participate in the study and for the processing of personal data.

Exclusion Criteria:

1. Recent (i.e. within the last 6 months) history of life-threatening asthma exacerbations;
2. Diagnosis of chronic obstructive pulmonary disease (COPD);
3. Asthmatic patients on treatment with biologic agents (e.g. monoclonal antibodies) and/or extemporary or fixed triple combinations (e.g. long-acting β2 agonist (LABA)/long-acting muscarinic antagonist (LAMA)/inhaled corticosteroid (ICS) at any dose regimen;
4. Patients with uncontrolled/clinically significant diseases (according to clinician's judgement) or inability to understand and fill in study questionnaires;
5. Concomitant participation in experimental clinical studies/investigations or participation in experimental clinical studies/investigations within 3 months prior to enrolment into the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Not adequately controlled asthmatic adult patients (according to clinician's judgement)
Sampling Method: Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Improvement of asthma control level using the 5-item Asthma Control Questionnaire | 6-month
  Proportion of patients improving the level of asthma control (based on ACQ-5 score).
  The ACQ-5 includes a measure of the top 5 asthma symptoms (woken at night by symptoms, day-time symptoms, limitation of daily activities, shortness of breath and wheeze) and the use of quick-relief bronchodilators.
  Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom and use questions on a 7-point scale (0 = no impairment, 6 = maximum impairment). Patients' scores are then classified into three groups ('grouped scores') as having well-controlled asthma (ACQ-5 score ≤0.75); not well-controlled nor poorly controlled asthma (ACQ-5 score 0.75-1.5), or poorly controlled asthma (ACQ-5 score ≥1.5)

SECONDARY OUTCOMES:
Improvement of asthma control level using the 5-item Asthma Control Questionnaire | 3 months
  Proportion of patients improving the level of asthma control (based on ACQ-5 score)
Achievement of minimal clinically important improvement in ACQ-5 score | 6 months
  Proportion of patients achieving minimal clinically important improvement in ACQ-5 scores, as defined by ACQ-5 score decrease of at least 0.5 points
Assessment of quality of life using EuroQol 5-dimension 5-level version (EQ-5D-5L) | 3 and 6 months
  Change in EQ-5D-5L score. It consists of 2 pages, a descriptive system and a visual Analogue scale. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each dimension having 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.The VAS records the respondent's self-rated health on a 10 cm vertical VAS with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
Assessment of adherence to treatment using 12-item Test of Adherence to Inhalers (TAI-12) | 3 and 6 months
  Change in TAI-12 score. TAI comprises a patient domain (including 10 items) and a healthcare professional domain (including 2 items). Each item ranges from 1 (lowest adherence) to 5 (highest adherence) points. The patient domain score ranges from 10 to 50. Adherence is rated as good (score =50), intermediate (score = 46-49), or poor (score ≤45). The questions for healthcare professionals are scored with 1 or 2 points (poor or good knowledge of the regimen and/or inhalation technique).
Structured questions on patient satisfaction about the inhaler | 3 and 6 months
  Three questions related to the satisfaction for the device will be administered to patients who will express the grade of agreement.
  The 3 questions are scored on a 0-4 Likert scale, which range from 0 (completely unsatisfied) to 4 (completely satisfied), for a total maximum score of 12. Higher scores indicate a higher satisfaction with the inhaler.
Asthma exacerbations | 6 months
  Occurrence of moderate-to-severe exacerbations
Adverse events | 6 months
  Number of AEs
Adverse drug reactions to BDP/FF NEXThaler | 6 months
  Number of ADRs

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale dell'Angelo, Mestre, VE, Italy

IPD SHARING:
Plan to Share IPD: No